CLINICAL TRIAL: NCT06253754
Title: Cerebral Hemodynamics and Cerebrospinal Fluid Dynamics in Postdural Puncture Headache An MRI Study for Exploring the Pathophysiological Mechanisms and Implication of Treatment
Brief Title: Pathophysiological Mechanisms and Implication of Treatment in Postural Puncture Headache
Acronym: PDPH
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-06754-01
Record Dates: First submitted 2024-02-01; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Post-Dural Puncture Headache
Keywords: MRI; Cerebral blood flow; Cerebrospinal fluid
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postdural puncture headache after lumbar puncture: Group of patients with aged 20-40 years undergoing planned neurological work-up including a lumbar puncture (LP). The group will include 40 subjects with and 40 subjects without PDPH.
  Interventions: Other: MRI examination
- Postdural puncture headache after accidental dural puncture: Group of parturients with EDA. The group will include 40 subjects with accidental dural puncture (ADP) with PDPH and 40 subjects without ADP and PDPH.
  Interventions: Other: MRI examination

INTERVENTIONS:
Other: MRI examination — All included subjects will be examined with MRI

SUMMARY:
To improve treatment for post dural puncture headache, its pathophysiology needs to be explored. Dural puncture alters CNS dynamics; using advanced MRI, we aim to investigate PDPHs pathophysiology explained by brain movement, cerebral blood flow, CSF dynamics and the effect of epidural blood patch.

DETAILED DESCRIPTION:
Post dural puncture headache (PDPH) is an iatrogenic and most common serious complication that can occur after a lumbar puncture or accidental dural puncture (ADP), as is often the case in women receiving epidural analgesia (EDA) during labour.

It is linked to substantial distress for patients specially mothers during the postpartum period, resulting in difficulties in forming a satisfying emotional bond with their newborns.

PDPH is a clinical diagnosis, based on symptoms and chronology of events and is therefore subjective since it relies on the patients' descriptions of symptoms and the clinician's interpretation of those symptoms.

Despite the lack of clear understanding of the pathophysiology of PDPH, several treatments have been suggested where an epidural blood patch (EBP) is considered the most effective option. Even though application of an EBP carries risks, symptom-relief is almost instantaneous, and the treatment has been shown to shorten hospital stay.

However, to improve treatment of these patients, a better understanding of its pathophysiology is needed to understand this condition more clearly. Even though PDPH is classified as a low-pressure headache it has been shown that the presence of PDPH does not always relate to a low CSF pressure nor does a normal pressure exclude PDPH. Our hypothesis is that the dural puncture, and the resulting outflow of CSF, changes intracerebral hemodynamics and dynamics of the CSF in a way that has never been fully investigated and described. Using magnet resonance imaging (MRI), including 4D phase contrast MRI it will be possible to quantify changes in hemodynamics and CSF dynamics in a new manner.

The main objective of this study is therefore to investigate the effects of dural puncture on cerebral blood flow (CBF) and cerebrospinal fluid (CSF) volume and pulsation and their relation to PDPH. This project will help to better understand the pathophysiology of PDPH and pave the way for improved management strategies in the future.

ELIGIBILITY:
Inclusion Criteria:

Postural puncture headache Age 20-40

Exclusion Criteria:

* Other central neurological disorders except the actual
* Acute medical condition
* Pregnancy
* Pacemaker, or other medical implants that are not MRI-compatible
* Invasive procedures on the central nervous system or surgery on the spine or brain in the last 12 months.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Two different study population with PDPH and controls.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-12-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Changes in cerebral dynamics with MRI | After 3 months
  Cerebral blood flow and CSF

CONTACTS AND LOCATIONS:
Overall Officials: Laleh Zarrinkoob, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Västerbotten County, Sweden